CLINICAL TRIAL: NCT00057759
Title: Treatment Of Erectile Dysfunction In Patients Treated On RTOG-9910 For Prostate Cancer: Impact On Patient And Partner Quality Of Life
Brief Title: Sildenafil in Treating Erectile Dysfunction in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RTOG-0215; CDR0000269135; NCI-P-02-0234; NCT00075127 (obsolete NCT alias)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Radiation Toxicity; Sexual Dysfunction; Sexuality and Reproductive Issues
Keywords: sexual dysfunction; sexuality and reproductive issues; radiation toxicity; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries; Sexual Dysfunction, Physiological; Sexuality | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil citrate (Experimental): Sildenafil with dose escalation as needed from 50 mg to 100 mg/day prn for 12 weeks.
  Interventions: Drug: sildenafil citrate
- Placebo (Placebo Comparator): Placebo with similar "dose escalation" opportunity for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: sildenafil citrate
  Arms: Sildenafil citrate
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Sildenafil may be effective in helping patients who have undergone treatment for prostate cancer to have an erection for sexual activity and may improve sexual satisfaction and quality of life.

PURPOSE: Randomized clinical trial to study the effectiveness of sildenafil in treating erectile dysfunction in patients who have undergone radiation therapy and hormone therapy for prostate cancer in clinical trial RTOG-9910.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of sildenafil vs placebo on erectile dysfunction in patients with prostate cancer treated with radiotherapy and antiandrogens on RTOG-9910.
* Compare the overall sexual function and satisfaction of patients treated with these regimens.
* Compare sexual satisfaction of partners of patients treated with these regimens.
* Compare patient and partner marital adjustment after treatment with these regimens.
* Determine factors that may predict response to sildenafil, including age, pretreatment sexual function, tobacco use, and comorbidities in these patients.

OUTLINE: This is a randomized, placebo-controlled, multicenter study. Patients are stratified according to prior use of sildenafil after treatment on RTOG-9910 and level of response (No vs yes [unsatisfactory] vs yes [satisfactory]), International Index of Erectile Function (IIEF) Question #1 score (0-1 vs 2-3), and RTOG-9910 treatment arm (I vs II). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sildenafil 1 hour prior to desired sexual intercourse.
* Arm II: Patients receive oral placebo 1 hour prior to desired sexual intercourse.

Treatment on both arms continues for 12 weeks. Patients then cross over to treatment on the other arm for 12 weeks.

Quality of life, including sexual function, marital adjustment, and partner's satisfaction, is assessed at baseline, at 12 and 25 weeks, and at 1 year.

Patients are followed at 1 year.

PROJECTED ACCRUAL: A total of 332 patients (166 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior treatment on RTOG-9910 for intermediate relapse-risk stage II or III prostate cancer as determined by any of the following combinations of factors:

  * T1b-4, Gleason score 2-6, and prostate-specific antigen (PSA) greater than 10 ng/mL but no greater than 100 ng/mL
  * T1b-4, Gleason score 7, and PSA less than 20 ng/mL
  * T1b-1c, Gleason score 8-10, and PSA less than 20 ng/mL
* Radiotherapy completed within the past 6 months to 5 years
* Pretreatment (before enrollment on this study) erectile dysfunction as measured by International Index of Erectile Function Question #1

  * Erectile dysfunction before starting prostate cancer therapy allowed
* Patients without partners or without partners willing to participate allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No myocardial infarction within the past year

Other

* No other invasive cancer within the past 5 years except localized basal cell or squamous cell skin cancer (stage 0-II)
* No anatomical genital abnormalities or concurrent conditions that would prohibit sexual intercourse or preclude study participation
* No other major medical or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 6 months since prior androgen suppression (e.g., leuprolide or goserelin), antiandrogen (e.g., bicalutamide, flutamide, or nilutamide), or estrogenic (e.g., diethylstilbestrol) agents

Radiotherapy

* See Disease Characteristics

Surgery

* No prior penile implant
* No prior bilateral orchiectomy

Other

* No concurrent sildenafil
* No concurrent participation in another medical research study to treat prostate cancer
* No concurrent organic nitrate or requirement for nitrates (e.g., nitroglycerin as needed)
* No concurrent ketoconazole, itraconazole, or erythromycin
* No concurrent use of mechanical (vacuum) devices or intracorporeal, intraurethral, topical, or oral agents for erectile dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Ability to obtain an erection, as measured by question 1 on the IIEF | From baseline to 12 weeks from the start of drug after crossover

SECONDARY OUTCOMES:
Overall sexual function and satisfaction as measured by the Sexual Adjustment Questionnaire (SAQ) | From baseline to 12 weeks from the start of drug after crossover
Partner sexual satisfaction as measured by the SAQ-Partner | From baseline to 12 weeks from the start of drug after crossover
Patient and spouse marital adjustment as measured by the Locke's Marital Adjustment Test | From baseline to 12 weeks from the start of drug after crossover
Predictors of erectile dysfunction therapy | From baseline to 12 weeks from the start of drug after crossover

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watkins Bruner, RN, PhD, Study Chair — Fox Chase Cancer Center
Locations (30):
- United States (30):
  - Mount Diablo Regional Cancer Center, Concord, California
  - Cancer Care Consultants Medical Associates at Daniel Freeman Memorial Hospital, Inglewood, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Cape Cod Hospital, Hyannis, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Community Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Akron City Hospital, Akron, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - LDS Hospital, Salt Lake City, Utah
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin

REFERENCES:
- [Result] Hanisch LJ, Bryan CJ, James JL, Pisansky TM, Corbett TB, Parliament MB, Stewart CE, Hartford AC, Sandler H, Berk LB, Kachnic L, Bruner DW. Impact of sildenafil on marital and sexual adjustment in patients and their wives after radiotherapy and short-term androgen suppression for prostate cancer: analysis of RTOG 0215. Support Care Cancer. 2012 Nov;20(11):2845-50. doi: 10.1007/s00520-012-1409-8. Epub 2012 Feb 22. PMID 22354624
- [Result] Watkins Bruner D, James JL, Bryan CJ, Pisansky TM, Rotman M, Corbett T, Speight J, Byhardt R, Sandler H, Bentzen S, Kachnic L, Berk L. Randomized, double-blinded, placebo-controlled crossover trial of treating erectile dysfunction with sildenafil after radiotherapy and short-term androgen deprivation therapy: results of RTOG 0215. J Sex Med. 2011 Apr;8(4):1228-38. doi: 10.1111/j.1743-6109.2010.02164.x. Epub 2011 Jan 14. PMID 21235716
- [Result] Bruner DW, James J, Pisansky TM, et al.: RTOG 0215 treatment of erectile dysfunction (ED) in patients treated with neoadjuvant and concurrent androgen deprivation (AD) and radiotherapy (RT) for prostate cancer (PC). [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-52, S30, 2007.